CLINICAL TRIAL: NCT03618992
Title: Improving the Appearance of Skin and Hair in Patients Undergoing Valley Fever Treatment
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator left university
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 1806645760
Record Dates: First submitted 2018-07-17; First posted 2018-08-07 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: Valley Fever; Coccidioidomycosis
Keywords: Valley Fever; Coccidioidomycosis
MeSH Terms: conditions — Coccidioidomycosis

STUDY DESIGN:
Intervention Model Description: Randomized control split body study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Active Comparator): Subjects will be provided with containers of topical cholesterol-containing moisturizers to be applied to the skin and hair, identical except for labels designating left and right. Topical formulations will be purchased by Skin Actives Scientific (www.skinactives.com), and will consist of one container of intervention and one of vehicle only (see ingredients below), to be applied to the left or right arm as indicated by pre-randomization assignment. Patients will be instructed to begin a 1-week washout period in which they will stop all topicals, and will then begin daily application of the topical intervention products to the indicated sites. Patients will return for follow-up visits at 2, 6, 10, and 14 weeks after starting intervention.
  Interventions: Other: Cholesterol-containing moisturizers
- Cohort 2 (No Intervention): Pre-study randomization will assign patients to have measurements obtained from either the left or right side of the body. Baseline skin barrier measurements of the skin and lips will be obtained, including transepidermal water loss (TEWL), hydration, pH and sebum (oil). Photos of the skin, lips, eyebrows, eyelashes and scalp will be taken. On each side, samples of scalp (pluck 1), eyebrow (trim 1), and eyelash (trim 1) hairs will be obtained only at baseline and the final visit. Patients will return for follow-up visits at 1, 2, and 3 months after discontinuation of oral antifungal therapy.
- Cohort 3 (No Intervention): Pre-study randomization will assign patients to have measurements obtained from either the left or right side of the body. Baseline skin barrier measurements of the skin and lips will be obtained, including transepidermal water loss (TEWL), hydration, pH and sebum (oil). Photos of the skin, lips, eyebrows, eyelashes and scalp will be taken. On each side of the body, samples of scalp (pluck 1, trim 1), eyebrow (pluck 1, trim 1), and eyelash (trim 1) hairs will be obtained at the baseline and final visit. Patients will return for follow-up visits at monthly intervals after initiation of oral antifungal therapy for up to 12 months.

INTERVENTIONS:
Other: Cholesterol-containing moisturizers — Commercially-available cholesterol containing topical formulations to be applied daily to the scalp, skin, lips, eyelashes, and eyebrows. Available from Skin Actives Scientific (www.skinactives.com).
  Arms: Cohort 1

SUMMARY:
This will be a multi-visit study that will take approximately 3 hours in total. Up to 200 subjects from the BUMC Valley Fever and BUMC Dermatology clinics will be enrolled in this study and assigned to one of three cohorts according to timeline of oral anti-fungal therapy. Subjects in Cohort 1 will be randomized to apply topical cholesterol-containing moisturizers to the skin, hair and lips on either the right or left side of the body daily. Measurements of skin barrier function, appearance of skin and hair, and hair samples will be obtained at baseline and at 4 week follow-up visits. Cohorts 2 and 3 will be observational groups at differing points in oral antifungal treatment regimen. Subjects will be randomized to have measurements of skin barrier function and hair and skin characteristics obtained from either the right or left side of the body at baseline and at monthly follow-up visits.

DETAILED DESCRIPTION:
Coccidioidomycosis, also known as Valley Fever, is a fungal condition most commonly seen in Arizona and can affect multiple organs, including the skin, lung, bone, joints, and central nervous system. Oral antifungal therapy such as fluconazole is the first-line medication to treat coccidioidomycosis. Through the investigator's clinical observations at the Valley Fever Center for Excellence, nearly all patients who have been placed on systemic azole treatment show some extent of cosmetic changes in their skin and hair, such as dry skin, chapped lips, hair loss, and change in hair characteristics. The goals of the study are to 1) understand the cosmetic changes in the skin and hair in patients initiating and discontinuing long-term oral antifungals, and 2) to examine whether cholesterol-based commercially-available moisturizers for the skin and for the hair can improve the cosmetic appearance better than a vehicle without these cholesterol ingredients.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, age 18 or older
* Patients who have been diagnosed with coccidioidomycosis (valley fever) requiring oral anti-fungal medications such as but not limited to fluconazoles
* Able to comprehend and read the English language

Exclusion Criteria:

* Subject does not fit inclusion criteria
* Children younger than 18 years of age
* Pregnant women
* Prisoners or those that are cognitively impaired
* Those with known allergies or intolerance to ingredients in the topical formulations
* Subject is unwilling or unable to comply with study procedures
* Unable to read or comprehend English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Skin barrier function - Transepidermal water loss (TEWL) | Up to one year
  Assess skin barrier function through measurement of transepidermal water loss (in g/m^2h) using a commercially-available, non-invasive device.
Skin barrier function - Stratum corneum hydration | Up to one year
  Assess skin barrier function through measurement of stratum corneum hydration (in arbitrary units) using a commercially-available, non-invasive device.
Skin barrier function - Sebum | Up to one year
  Assess skin barrier function through measurement of sebum (in micrograms/cm^2) using a commercially-available, non-invasive device.
Skin barrier function - pH | Up to one year
  Assess skin barrier function through measurement of stratum corneum pH (in pH units) using a commercially-available, non-invasive device.

OTHER OUTCOMES:
Hair characteristics | Up to one year
  Evaluate caliber and density of scalp, eyebrow and eyelash hair through hair samples and photos.

CONTACTS AND LOCATIONS:
Overall Officials: Vivian Shi, MD, Principal Investigator — University of Arizona
Locations (2):
- United States (2):
  - University of Arizona - Banner University Medicine Dermatology, Tucson, Arizona
  - Valley Fever Center for Excellence, Tucson, Arizona